CLINICAL TRIAL: NCT03627533
Title: The Differences of Oocyte Maturation, Granulosa Cell Apoptosis Index Between Electroacupuncture And Sham Groups IVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, nadia oktari, principal investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Medical Acupuncture
Record Dates: First submitted 2018-08-02; First posted 2018-08-13 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Acupuncture; in Vitro Fertilization; BCL2 Gene mRNA Overexpression; Oocyte Maturation
MeSH Terms: interventions — Electroacupuncture

STUDY DESIGN:
Intervention Model Description: electroacupuncture versus sham electroacupuncture
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture (Experimental): Electroacupuncture therapy is done at the point of CV3 Zhongji, CV4 Guanyuan, and EXCA-1 Zigong with continuous wave, 2 Hz frequency for 30 minutes. Acupuncture manuals on MA-IC3 endocrine (ear points), GV20 Baihui, ST36 Zusanli, SP6 Sanyinjiao, BL57 Chengsan and KI3 Taixi for 30 minutes.
  Interventions: Procedure: Electroacupuncture
- Sham electroacupuncture (Sham Comparator): Sham electroacupuncture are done at same electroacupuncture point location but puncture are not done, also electro stimulator are turned off.
  Interventions: Procedure: Electroacupuncture

INTERVENTIONS:
Procedure: Electroacupuncture — Electroacupuncture therapy is done at the point of CV3 Zhongji, CV4 Guanyuan, and EXCA-1 Zigong with continuous wave, 2 Hz frequency for 30 minutes. Acupuncture manuals on endocrine ear points, GV20 Baihui, ST36 Zusanli, SP6 Sanyinjiao, BL57 Chengsan and KI3 Taixi for 30 minutes.

SUMMARY:
Interventional studies compared electroacupuncture group versus sham electroacupuncture group to granulosa cell apoptosis index, oocyte maturation, GDF9 and BMP15 levels, and fertilization rate in in vitro fertilization program

DETAILED DESCRIPTION:
The study was conducted at the Dr.Cipto Mangunkusumo National General Hospital, Indonesia in September - November 2018.The inclusion criteria are patients who underwent controlled ovarian stimulation with antagonist protocol, age 30-39 years, BMI <29kg / m2. Exclusion criteria were not having a skin infection at acupuncture point and not using a pacemaker. Then patients were randomly divided into two groups: electroacupuncture and sham electroacupuncture. Electroacupuncture therapy was done 6 times at: 2 times before and 4 times during controlled ovarian stimulation.Apoptotic index of granulosa cells were examined by quantitative real time PCR techniques for BAX/BCL-2 expression.Oocyte maturation and fertilization rate output parameters are examined by competent embryologists after ovum pick up while GDF9 and BMP15 levels were examined by quantitative real time PCR techniques for GDF9 and BMP15 mRNA expression

ELIGIBILITY:
Inclusion Criteria:

* women underwent controlled ovarian stimulation with antagonist protocol
* BMI < 29 kg/m2
* willing and sign the inform consent
* follow the research until completed

Exclusion Criteria:

* having skin infection at acupoint location
* use a pacemaker

Ages: 30 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Index apoptotic (Ratio Bax/Bcl-2) of granulosa cells, GDF9 and BMP15 | "up to 1 months"
  Bax/Bcl-2 is proapoptotic protein compare to antiapoptotic protein. GDF9 and BMP15 protein expression

SECONDARY OUTCOMES:
oocyte maturation index | "up to 1 months"
  fertilization rate is number of fertilized oocytes compared with all total number oocyte which taken when ovum pick-up. oocyte maturation index is the number of mature oocyte (metaphase II oocyte) compare with all total number oocyte which taken when ovum pick-up
Fertilization rate | "up to 1 months"
  fertilization rate is number of fertilized oocytes compared with all total number oocyte which taken when ovum pick-up.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Simadibrata, MD, Study Chair — Medical Acupuncture of Indonesian University
Locations (1):
- Indonesian University, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No